CLINICAL TRIAL: NCT06213688
Title: The Impact of Pollutants on Patients With Psoriasis or Atopic Dermatitis by Investigating the Activation of the Aromatic Hydrocarbon Receptor.
Brief Title: Involvement of Pollutants in Atopic Dermatitis and Psoriasis
Acronym: DIAhR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: ALPHENYX (Unknown); Aix Marseille Université (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM23_0328
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: Atopic dermatitis; Psoriasis; Aryl hydrocarbon receptor; Dioxins; Polycyclic aromatic hydrocarbons; Pollution
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Other): Patients with atopic dermatitis or psoriasis
  Interventions: Other: blood sampling; Other: urine sampling
- Controls (Other): Patients have consulted or been hospitalized for dermatological reasons without psoriasis or atopic dermatitis
  Interventions: Other: blood sampling; Other: urine sampling

INTERVENTIONS:
Other: blood sampling — blood sampling at inclusion
Other: urine sampling — urine sampling at inclusion

SUMMARY:
Introduction Pollution is a significant public health issue. Research has shown a positive correlation between air pollution and chronic inflammatory dermatoses, including psoriasis and eczema. The incidence of these diseases has been steadily increasing since the beginning of industrialization. The mechanism behind this association involves the activation of the aromatic hydrocarbon receptor (AhR). The aryl hydrocarbon receptor (AhR) plays a role in regulating the balance between T helper 17 (TH17) and regulatory T cells (TREG), as well as in generating oxidative stress and producing pro-inflammatory cytokines. Studies in cultured keratinocytes have shown that a non-competitive antagonist that modulates AhR activity can reduce cutaneous inflammatory processes induced by polycyclic aromatic hydrocarbons (PAHs).

Objectives:

It has been suggested that activation of the AhR by PAHs and dioxins may be related to the pathogenesis of atopic dermatitis and psoriasis. The main objective is to compare the levels of AhR pathway activation markers between cases and controls. Secondary objectives include correlating environmental exposure to AhR ligands with disease severity in patients. Finally, we will compare the expression of inflammatory and AhR activation markers in cultured peripheral blood mononuclear cells (PBMCs) after in vitro stimulation with benzo(a)pyrene.

Material and methods:

The study will measure exposure to pollutants by determining blood dioxins and urinary PAH metabolites. Pro-inflammatory cytokines IL1β, TNFα, IL23, IL17 and IFNγ and Malondialdehyde (MDA) serum concentrations will be measured by ELISA. The TREG and TH17 lymphocyte population ratio will be evaluated by flow cytometry on isolated PBMCs. Additionally, the level of expression of CYP 1A1 and 1B1, pollutant-metabolizing enzymes induced by AhR, will be assessed on isolated PBMCs. The expression levels of the AhR and NfkB active fractions will be determined by immunofluorescence. Subsequently, levels of AhR activation markers will be compared after stimulation of PBMCs with benzo(a)pyrene.

DETAILED DESCRIPTION:
I. Introduction Pollution is a significant component of the exposome, with established links to human health. In 2019, pollution was estimated to be responsible for 9 million premature deaths, making it the fourth leading risk factor for mortality worldwide. Over the last 20 years, pollution-related deaths have increased by 66%. This is due to industrialization, uncontrolled urbanization, population growth, burning fossil fuels, and a lack of restrictive policies in some regions.

The cutaneous layer is composed of a complex network of cells that form a mechanical and biological barrier essential for maintaining the body's integrity and homeostasis. Pollution can directly impair this function by crossing the barrier or entering the systemic circulation through inhalation or ingestion.

Atopic dermatitis (AD) and psoriasis are chronic inflammatory skin conditions with multifactorial origins, including genetic predisposition, immune dysregulation, and environmental factors. Epidemiological studies have shown a positive correlation between air pollution and the development of these diseases.

Given their high prevalence and the impact of symptoms on patients' quality of life, a better understanding of the exposome in these diseases represents a major challenge.

Experimental studies have demonstrated that the aromatic hydrocarbon receptor (AhR) pathway plays a significant role in the impact of pollutants on psoriasis and AD. AhR is a transcription factor involved in the response to environmental pollutants, which remains inactive in a cytoplasmic complex with chaperone proteins. Upon binding with its ligand, AhR translocates to the nucleus and dimerizes with its nuclear partner, Arnt. The activation of the complex leads to the expression of numerous genes that contain a consensus sequence known as the xenobiotic response element (XRE) in their promoters.

The activator ligands of the AhR comprise xenobiotics found in the environment, primarily polycyclic aromatic hydrocarbons (PAHs), dioxins, and so-called 'dioxin-like' compounds 12. This signalling pathway is considered an 'adaptive' response to detoxify the body from various exogenous compounds. However, prolonged activation of the AhR by such agents may lead to deregulation of the inflammatory process, contributing to the development of psoriasis and AD.

The aryl hydrocarbon receptor (AhR) regulates the transcription of cytochromes 1A1 (CYP1A1) and 1B1 (CYP1B1), which are members of a multigene family of enzymes involved in xenobiotic metabolism. These enzymes catalyse the bioactivation of HAPs into electrophilic metabolites leading to activation of NFκB, a key player in the inflammatory response. During their catalytic cycle, these CYP1 enzymes produce reactive oxygen species (ROS), which generate oxidative stress. In addition, the AhR is responsible for regulating the expression of pro-inflammatory cytokines, including IL1β, TNFα, IL23, IL17 and IFNγ. It can directly affect the balance between Th17 lymphocytes and regulatory T cells (Tregs), potentially contributing to cutaneous inflammatory processes.

However, further research is needed to better define the role of AhR in the pathogenesis of chronic inflammatory dermatoses. This will help in the management and prevention of these diseases, especially when environmental risk factors are associated with predisposition.

II. Objective:

It is hypothesized that the activation of AhR with exogenous ligands may play a role in the development of atopic dermatitis and psoriasis.

The main objective is to compare the levels of AhR pathway activation markers between cases and controls.

Secondary objectives include correlating environmental exposure to AhR ligands with disease severity in patients.

Finally, we will compare the expression of inflammatory and AhR activation markers in cultured peripheral blood mononuclear cells (PBMCs) after in vitro stimulation with benzo(a)pyrene.

III. Material and methods:

We will be carrying out a case-control study:

* Case: Patients with chronic inflammatory dermatosis corresponding to psoriasis or atopic dermatitis.
* Controls: People consulting the dermatology department who do not have these pathologies.

All participants, including patients and controls, will undergo consultation/hospitalisation and biological testing as part of their usual medical care. Procedures performed as part of the protocol will not interfere with their care.

A sample of 10 ml of blood will be taken for toxicological analysis. 20 ml of blood will be taken for evaluation of inflammatory and AhR activation markers.

A. Pollutant measurement The blood sample will be centrifuged, the serum will then be collected and stored at -20 C until the blood dioxins are analysed. 2,3,7,8-tétrachlorodibenzo-p-dioxin (TCDD) and polychlorobiphényle 118 (PCB118) will be measured in blood using gas chromatography coupled with high-resolution mass spectrometry (GC-HR-MS).

For biological monitoring of exposure to PAHs,1-Hydroxypyrene (1-OHP) will be measured in urine using high-performance liquid chromatography-mass spectrometry (LC-MS-MS)

B. Evaluation of inflammatory and AhR activation markers

* PBMCs will be isolated from a 20mL blood sample using a standard Ficoll® gradient protocol. The isolated cells and sera will be aliquoted and frozen for subsequent experiments on the AhR signalling pathway.
* Enzyme-Linked Immunosorbent Assay (ELISA) will be used to measure pro-inflammatory cytokines IL1β, TNFα, IL23, IL17 and IFNγ.
* Malondialdehyde (MDA) concentration will be determined using the ELISA method as a biomarker for lipid peroxidation, which indicates the level of oxidative stress caused by reactive oxygen species (ROS).
* Fluorochrome-conjugated monoclonal antibodies (CD4, CD25, CD127, FOXP3, Il17) will be used in fluorescence activated cell sorter (FACS) to assess the numbers and ratios of different lymphocyte populations in PBMCs. The investigation will focus on Th17 and Treg levels.
* FACS will be used to assess the expression of CYP1A1 and CYP1B1, which are prototypes of AhR target genes, in PBMCs after specific targeting.
* The levels of expression of the active fractions of AhR and NfkB will be determined using direct immunofluorescence technique.
* PBMCs will be cultured with anti-CD3+/-BaP (50 nM) in a cell incubator (37°C, 5% CO2+ controlled humidity) for 48-72 hours. The parameters of interest, including oxidative stress, pro-inflammatory cytokines, and assessment of the AhR pathway, will be reassessed after lymphocyte reactivation by anti-CD3 in the presence or absence of BaP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85.
* The study's participants possess the capacity to comprehend the research.
* Patients have consulted or been hospitalized for dermatological reasons
* Patients undergo biological monitoring as part of their routine care.
* Having psoriasis or atopic dermatitis for more than 6 weeks (cases)
* Subjects with a PASI severity score (psoriasis) greater than 5 and an EASI score (atopic dermatitis) greater than 12 at inclusion (cases)

Exclusion Criteria:

* Active smoking or less than 3 months since quitting
* Pregnancy
* Biotherapy treatment in progress or in the 8 weeks prior to inclusion
* Immunotherapy treatment in progress or in the 6 months prior to inclusion
* Chemotherapy treatment in progress or in the 4 weeks prior to inclusion
* Person in an emergency situation, adult subject to a legal protection measure (adult under guardianship, curatorship or safeguard of justice).
* Non-affiliation with a social security scheme (beneficiary or dependent).
* Subjects with a history of autoimmune diseases (controls)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Determination of CYP 1A1/1B1 in PBMCs | Inclusion
  The expression of CYP1A1 and CYP1B1 in PBMCs in ng/mL is used as primary endpoint;

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marie-Aleth, Principal Investigator — AP-HM

IPD SHARING:
Plan to Share IPD: No